CLINICAL TRIAL: NCT02307916
Title: Fibroblast Growth Factor Regeneration of Tympanic Membrane Perforations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: D. Bradley Welling, MD, PhD (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, D. Bradley Welling, MD, PhD, Principal Investigator, M.D., Ph.D., Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-043
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Results first posted 2020-06-11 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2020-12

CONDITIONS: Tympanic Membrane Perforation
Keywords: tympanic membrane perforation; ear drum; hole
MeSH Terms: conditions — Tympanic Membrane Perforation | interventions — Fibroblast Growth Factor 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FGF-2 (Experimental): FGF-2 given a minimum of 1 and maximum of 3 times within, approximately, 60 days.
  Interventions: Drug: FGF-2
- Placebo (Placebo Comparator): Equal concentration of saline is given a minimum of 1 and maximum of 3 times within, approximately, 60 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: FGF-2 — The FGF-2 method of use comprises a pledget of gelatin foam with human fibroblast growth factor-2 (FGF-2) added to the pledget just before topical application to the tympanic membrane, and the use of Tisseel, a fibrin glue used for applications in ear surgery.
  Other Names: FGF2, Human Fibroblast Growth Factor 2
  Arms: FGF-2
Other: Placebo — Placebo comparator using a sterile saline solution.
  Other Names: Placebo comparator; sterile saline
  Arms: Placebo

SUMMARY:
A Phase II randomized trial will be initiated to evaluate closure of the perforated tympanic membrane as the primary measureable outcome. The goal is to determine the safety and efficacy of Fibroblast Growth Factor-2 (FGF-2) in the closure of chronic tympanic membrane perforations (TMP). If FGF-2 is topically applied for the treatment of chronic TMP in humans, it is hypothesized it will be safe, tolerable and effective for use as treatment for tympanic membrane perforation. A total of 60 subjects will be recruited.

DETAILED DESCRIPTION:
A Phase II randomized trial will be initiated to evaluate efficacy as the primary measureable outcome. Eligible and consented patients will be randomized in a 3:1 ratio to the optimal biologic dose (OBD) of FGF-2 or placebo (sterile water).

Application of the study treatment may occur at the initial Screening Visit (pending all eligibility requirements can be confirmed) or at Visit 1 and may be repeated at each follow up visit as needed for a maximum of three treatments per treatment arm. These follow up visits will occur three weeks (+/- 7 days) from the last treatment application. During these visits, the subject's tympanic membrane will be examined, photographed, and additional otologic tests will be performed. If the perforation is found to be closed during these visits, then the subject will report in 2 months (+/-7 days) for a final study visit.

If the subject's TMP has not closed after the third and final application of their assigned treatment group, then the subject will be crossed over to the other treatment group. Again, the subject may be given up to three additional treatments in this new group. The follow up visits will follow the same schedule, occurring three weeks (+/- 7 days) from the last treatment. The same otologic procedures will be performed as in the previous visits.

All subjects will report for a final study visit 2 months (+/- 7 days) after their last follow up visit when the perforation is determined to be closed or when the subject has completed the maximum number of study visits without perforation closure. The study will be completed for reporting purposes after all subjects have completed the 2 month (+/- 7 days) follow up final visit.

ELIGIBILITY:
Inclusion Criteria:

1. Dry tympanic membrane perforation of greater than 3 months duration
2. If female, post-menopausal or sterile, or if she is of child-bearing potential, must have a negative beta-human chorionic gonadotropin (HCG) test and must be using an adequate form of birth control such as birth control pills, birth control implants, intrauterine devices (IUDs), diaphragms or condoms.

Exclusion Criteria:

The presence of any of the following excludes a subject from study enrollment:

* Active otitis media or chronic otorrhea from the middle ear
* Subjects receiving radiation therapy, corticosteroids, immunosuppressive agents or chemotherapy
* Subjects who, at study entry, are taking systemic antibiotics
* Subjects who are immunosuppressed
* Subjects experiencing bacterial or viral infection or who may otherwise be febrile
* Life expectancy of less than 1 year
* Active alcohol or drug abuse within 6 months prior to study entry
* Significant medical condition that could prevent full participation in the procedures required for the study (See body of protocol for full list of exclusions)
* Known or suspected allergies to any components used in the study
* Subjects who have cholesteatoma mass in the tympanic cavity
* Subjects whose total perforation cannot be seen by an endoscope
* Subjects with inadequately controlled diabetes mellitus (NGSP: HbA1c 6.9% or higher)
* Subjects with a history of malignant ear canal tumors within 3 years of screening for eligibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-10; Primary Completion 2019-07 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D. B. Welling, M.D., Ph.D, Principal Investigator — Massachusetts Eye and Ear
Locations (2):
- United States (2):
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - Wilford Hall, Lackland Airforce Base, Lackland City, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who met exclusion criteria were considered "screen-fail" and were not assigned to a randomization group.
Period: Overall Study
Arm/Group | FGF-2 | Placebo
Started | 42 | 15
Completed | 40 | 14
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FGF-2 | Placebo | Total
Number analyzed (Participants) | 42 | 15 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 10 | 42
  >=65 years | 10 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (13.9) | 55.8 (15) | 52.7 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 8 | 31
  Male | 19 | 7 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 42 | 15 | 57

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Tympanic Membrane Closure Following Treatment
Description: The efficacy of the treatment is determined by the number of patients whose tympanic membrane perforations closed after study treatments. Subjects from both treatment arms received up to three treatments before determining non-closure of the tympanic membrane.
Time Frame: ~60 days
Measure: Count of Participants; unit: Participants
Arm/Group | FGF-2 | Placebo
Number analyzed (Participants) | 40 | 14
Participants | 23 | 10

2. Secondary Outcome: Measurement of Changes in Pure-tone Averages
Description: measured by pre- and post-treatment audiograms.
Time Frame: Baseline, 60 days
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | FGF-2 | Placebo
Number analyzed (Participants) | 40 | 14
dB | 7.9 (8.8) | 5.9 (9.1)

3. Secondary Outcome: Measurement of Changes in Speech Discrimination Scores
Description: Speech discrimination score is determined by having the patient listen to words through headphones and having the patient repeat the words back to the audiologist. A score of 100 percent (100%) is the best outcome, and 0 percent (0%) is the worst. Pre- and post- treatment tests are compared and analyzed.
Time Frame: Baseline, 60 days
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | FGF-2 | Placebo
Number analyzed (Participants) | 40 | 14
percent | 3.2 (8.1) | 1.7 (4.7)

4. Secondary Outcome: Number of Treatments Required for Closure of the Tympanic Membrane Perforation
Description: Out of the patients who healed, some healed with 1 treatment, some with 2 treatments, and some with 3 treatments.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: treatments
Arm/Group | FGF-2 | Placebo
Number analyzed (Participants) | 40 | 14
treatments | 1.4 (0.6) | 1.7 (0.6)

5. Secondary Outcome: Number of Patients With Normal Mobility of the Eardrum as Assessed by Tympanometry
Description: Tympanometry is an examination used to test the condition of the middle ear and the mobility of the eardrum. Any type of perforation, regardless of size, would cause the result of the tympanometry to be abnormal. We use this test to determine if the eardrum closed completely.
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | FGF-2 | Placebo
Number analyzed (Participants) | 40 | 14
Participants | 23 | 10

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of enrollment to the final follow-up visit, usually within 6 months.
Arm/Group | FGF-2 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/15
Other Adverse Events (participants affected / at risk) | 13/42 | 5/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FGF-2 (N=42) | Placebo (N=15)
Ear drainage post-treatment (Ear and labyrinth disorders) | 5 (9) | 2 (2)
Ear pain during procedure (Ear and labyrinth disorders) | 3 (3) | 2 (4)
Ear infection (Ear and labyrinth disorders) | 5 (7) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-28): https://cdn.clinicaltrials.gov/large-docs/16/NCT02307916/Prot_SAP_000.pdf